CLINICAL TRIAL: NCT04198454
Title: Randomized, Investigator-blinded Study of Compression in Wound Healing With and Without Fractional Ablative CO2 Laser After Excisions on the Lower Extremity (CHIME+)
Brief Title: Compression and CO2 Laser for Leg Wounds
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: STU00211239
Record Dates: First submitted 2019-12-12; First posted 2019-12-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Wound Healing
MeSH Terms: interventions — Compression Bandages

STUDY DESIGN:
Intervention Model Description: Sequential, multiple assignment, randomized trials (SMARTs)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Compression bandages (Active Comparator): Class I (20-30 mmHg) compression bandages or stocking. This is considered a standard measure in the recovery of lower extremity wounds and often recommended.
  Interventions: Other: Compression bandages
- Standard wound dressings (Other): Wound dressings alone consisting of gauze and skin tape to cover the wound.
  Interventions: Other: Standard wound dressings
- Compression bandages with FACL (Experimental): Class I compression (20-30 mmHg) bandage or stocking with FACL.
  Interventions: Other: Compression bandages; Device: Fractional ablative carbon dioxide laser

INTERVENTIONS:
Other: Compression bandages — Class I (20-30 mmHg) compression bandages or stocking
  Arms: Compression bandages; Compression bandages with FACL
Other: Standard wound dressings — Wound dressings alone consisting of gauze and skin tape to cover the wound
  Arms: Standard wound dressings
Device: Fractional ablative carbon dioxide laser — Participant will have laser applied to their wound bed.
  Arms: Compression bandages with FACL

SUMMARY:
The purpose of this study is to determine the efficacy and safety of compression bandaging with fractional ablative carbon dioxide laser (FACL) compared to compression and standard dressings alone for healing of post-operative wounds of the leg.

This is a randomized, SMART design, clinical trial. Approximately 80 participants will be randomized to initially receive compression bandages or standard wound dressings after surgery on the lower leg. After 4 weeks, the group assigned to compression bandages will be further randomized to either continue with the compression bandages only or continue with the compression bandages and also receive (FACL). The study is designed as an 6-month study. This study was a pilot study designed to determine feasibility of these procedure.

Subjects currently living in the Chicago metropolitan area and meet inclusion/exclusion criteria will be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:Patients will be identified through the clinic where their skin is to be treated by excisional surgery on the lower leg. Those considered for enrollment must also meet the following criteria:

1. >18 years of age
2. Wound size of at least 1 cm in width
3. Cutaneous excision of the lower leg
4. Surgeon elected repair of healing by secondary intention
5. Participants must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

1. Current smoker
2. Uncontrolled diabetes mellitus
3. Uncontrolled hypothyroidism
4. Severe renal impairment or hypoalbuminemia
5. Chronic lymphedema
6. Severe venous insufficiency (large varicose veins, atrophie blanche)
7. Arterial insufficiency (ABI < 0.8)
8. Rubber or rubber accelerator allergy
9. Prior radiation to the surgical site
10. History or evidence of a clinically significant medical or psychiatric disorder, condition or disease that in the opinion of the treating physician would pose a risk or interfere with evaluation or completion of the study
11. Subject un willing to sign an IRB approved consent form
12. Participants who are unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-02-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mean change wound size as determined by measurements | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No